CLINICAL TRIAL: NCT01999309
Title: Simvastatin Addition for Patients With Recent-onset Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iris Sommer (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, Iris Sommer, Prof. Dr., UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43806
Record Dates: First submitted 2013-11-14; First posted 2013-12-03 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Psychosis NOS
Keywords: Schizophrenia spectrum disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Experimental): The lipid-lowering drug simvastatin is added to normal antipsychotic treatment. One 40 mg simvastatin tablet daily for the treatment period of one year.
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Placebo is added to normal antipsychotic treatment. One identical looking placebo tablet daily for the treatment period of one year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — The lipid-lowering drug simvastatin is added to normal antipsychotic treatment. One 40 mg simvastatin tablet daily for the treatment period of one year.
  Other Names: Zocor
  Arms: Simvastatin
Drug: Placebo — Placebo is added to normal antipsychotic treatment. One identical looking placebo tablet daily for the treatment period of one year.
  Arms: Placebo

SUMMARY:
Rationale: There is ample evidence that inflammatory processes play a role in the pathophysiology of schizophrenia. Although Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) have been shown to be able to reduce symptoms in these patients, these drugs either have unfavourable cardiovascular side effects or are otherwise not well tolerated. Moreover, patients with schizophrenia already tend to have an increased cardiovascular risk. The combination of well-established vascular protection and reduction of inflammation by simvastatin offers a highly attractive potential to further improve the treatment of schizophrenia and related disorders.

Hypotheses: Daily treatment with 40mg simvastatin in addition to antipsychotic treatment reduces psychotic symptoms, improves cognition, attenuates brain volume loss, and decreases the risk for metabolic syndrome as well as for movement disorders, when compared to placebo.

Objective: The primary objective of this trial is to investigate the proposed beneficial effect of simvastatin as compared to placebo when given for one year in addition to antipsychotic medication to patients with psychotic disorder. We expect lower symptom severity as measured with the PANSS (Positive and Negative Syndrome Scale) and less cognitive decline as measured with the BACS (Brief Assessment of Cognition in Schizophrenia).Secondary objectives are assessment of general functioning, presence and severity of metabolic syndrome and degree of movement disorders, and assessments of brain volume. Lastly, we examine various immunological parameters in serum and peripheral blood mononuclear cells and the experience of childhood trauma.

Study design: Randomized placebo-controlled double-blind trial.

Study population: 150 men and women, between 18 and 50 years of age, diagnosed with schizophrenia, schizoaffective or schizophreniform disorder (DSM-IV 295.*) or psychosis NOS (not otherwise specified) (298.9). Onset of first psychosis no longer than 3 years ago.

Intervention: Patients will be randomized 1:1 to either 40 mg simvastatin or placebo daily, in the form of identical tablets.

DETAILED DESCRIPTION:
Rationale: Different lines of evidence now suggest that low grade inflammation in the central nervous system is involved in the pathogenesis of schizophrenia. These include the altered risk of schizophrenia patients and their relatives for specific auto-immune diseases, clinical similarities between the course of schizophrenia and auto-immune disease and decreased prevalence of schizophrenia in men who have used Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) or glucocorticosteroids for somatic disorders. Furthermore, an infectious cause or trigger is suggested by the observed association between schizophrenia and pre- and perinatal infections, as well as by seroconversion to certain pathogens in patients with schizophrenia. On a cellular level, inflammation of the central nervous system is suggested by an increased number of activated microglia cells in the brains of patients with schizophrenia as visualized by positron electron tomography. In an activated state, microglia cells can produce free radicals, pro-inflammatory components and other neurotoxic substances, causing cell death in their proximity. The activation of microglia cells provides a possible route by which an increased pro-inflammatory state in the brain could cause increased gray matter loss and more severe negative and cognitive symptoms. Although Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) have been shown to be able to reduce symptoms in these patients, these drugs either have unfavourable cardiovascular side effects or are otherwise not well tolerated. Moreover, patients with schizophrenia already tend to have an increased cardiovascular risk. The combination of well-established vascular protection and reduction of inflammation by simvastatin offers a highly attractive potential to further improve the treatment of schizophrenia and related disorders.

Hypotheses: Daily treatment with 40mg simvastatin in addition to antipsychotic treatment reduces psychotic symptoms, improves cognition, attenuates brain volume loss, and decreases the risk for metabolic syndrome as well as for movement disorders, when compared to placebo.

Objective: The primary objective of this trial is to investigate the proposed beneficial effect of simvastatin as compared to placebo when given for one year in addition to antipsychotic medication to patients with psychotic disorder. We expect lower symptom severity as measured with the Positive And Negative Symptom Scale (PANSS) and less cognitive decline as measured with the Brief Assessment of Cognition in Schizophrenia (BACS).Secondary objectives are assessment of general functioning using the General Assessment of Functioning (GAF), presence and severity of metabolic syndrome, as defined by the American Heart Association/National Heart, Lung and Blood Institute (AHA/NHLB), presence and severity of movement disorders using validated scales, and assessments of brain volume through magnetic resonance imaging (MRI). Lastly, we examine various immunological parameters in serum and peripheral blood mononuclear cells and the experience of childhood trauma using the Childhood Trauma Questionnaire Short Form (CTQ-SF).

Study design: Randomized placebo-controlled double-blind trial.

Study population: 150 men and women, between 18 and 50 years of age, diagnosed with schizophrenia, schizoaffective or schizophreniform disorder (DSM-IV 295.*) or psychosis NOS (not otherwise specified) (298.9). Duration of disease should be no more than three years.

Intervention: Patients will be randomized 1:1 to either 40 mg simvastatin or placebo daily, in the form of identical tablets.

Main study parameters/endpoints: Primary outcome is change in total symptom severity (PANSS score) from baseline to end of treatment. Secondary outcomes will be the changes in GAF scores, cognitive functioning, presence and severity of metabolic syndrome and movement disorders and assessment of brain volume change, in addition to the measurement of various immunological biomarkers, childhood trauma. and depression symptoms.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Use of simvastatin implies that there is a risk of side effects, as all lipid-lowering drugs carry the risk of negative effects. The number of patient visits will be limited and mainly requires time investment for a few physical examinations, questionnaires and two cognitive testing sessions (around 10 hours per year in total).

Blood will be drawn at four occasions with negligible and known risks (e.g. irritation). The burden and risks are acceptable while the benefits are expected to be considerable.

ELIGIBILITY:
Inclusion Criteria:

* A DSM-IV-R diagnosis of: 295.x (schizophrenia, schizophreniform disorder, or schizoaffective disorder) or 298.9 (psychosis NOS)
* Onset of first psychosis no longer than 3 years ago.
* Age between 18 and 50 years
* Written informed consent is obtained
* Female patients of childbearing potential need to utilize a proper method of contraception (the pill, vaginal ring, hormonal patch, intrauterine device, cervical cape, condom, contraceptive injection, diaphragm) in case of sexual intercourse during the study.

Exclusion Criteria:

* Fulfilment of criteria for statin prescription; according to the Dutch Heart Foundation, statin treatment is indicated when the total cholesterol level is > 8 mmol/l (www.hartstichting.nl)
* Presence of any of the contra-indications or warnings for the use of simvastatin as reported in the SPC (Summary of Product Characteristics)
* Chronic use of glucocorticosteroids (temporary use is permitted, if stopped at least 1 month before start of treatment trial)
* Chronic use of non-steroidal anti-inflammatory drugs (temporary use is permitted, if stopped at least 1 month before start of treatment trial)
* Current use of statins or other lipid-lowering drugs
* Pregnancy or breast-feeding
* Active liver, kidney or muscle disease as defined by alanine aminotransferase (ALAT), creatinine or creatine kinase (CK) levels more than two times the upper boundary of normal levels
* In case of familial risk for muscular disorders or previously experienced muscle toxicity when taking medication similar to simvastatin, creatine kinase (CK) levels will also be checked (as recommended by the Dutch Farmacotherapeutisch Kompas, www.farmacotherapeutischkompas.nl/). In addition, levels of aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), gammaglutamyltranspeptidase (γ-GT) and creatinine will be checked when a history of alcohol abuse, liver or kidney disorders is reported.
* Use of comedication that either inhibits or induces the live enzyme CYP3A4 which is responsible for the degradation of simvastatin. Inhibitors of CYP3A4 include itraconazole, ketoconazole, posaconazole, fluconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, nefazodone, telaprevir, boceprevir, imatinib, ticagrelor, voriconazole; inducers of CYP3A4 include carbamazepin, efavirenz, nevirapine, etravirine (can be washed out before start of trial)
* Use of comedication that may increase the risk for myalgia, rhabdomyolysis and myopathy, including colchicine, bosentan, phenobarbital, phenytoin, hypericum, rifabutin, rifampicin, fibrates (e.g. gemfibrozil), fusidic acid, carbamazepin (can be washed out before start of trial)

For patients, the MRI scan requires addition exclusion criteria to be eligible to participate in this part of the study (if these additional criteria are not met, patients can participate in the study but not in the MRI component):

* Ferrous objects in or around the body (e.g. braces, glasses, pacemaker, metal fragments)
* Claustrophobia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Total symptom severity | 0, 1, 3, 6, 9 and 12 months
  Change in Positive And Negative Syndrome Scale (PANSS) total score

SECONDARY OUTCOMES:
Change in positive, negative and general symptom severity | 0, 1, 3, 6, 9 and 12 months
  Change in PANSS positive, negative and general psychopathology scale scores
Global functioning | 0, 1, 3, 6, 9, and 12 months
  Change in Global Assessment of functioning scale (GAF) score
Change in cognitive functioning | 0 and 12 months
  Total score of the Brief Assessment of Cognition in Schizophrenia (BACS)
Presence and severity of metabolic syndrome | 0, 1, 6 and 12 months
  As defined by the American Heart Association/National Heart, Lung and Blood Institute. The definitions and reference ranges for metabolic syndrome are:
  * Abdominal obesity (waist circumference) men ≥ 102 cm, women ≥ 88 cm
  * Triglycerides ≥ 150 mg/dL
  * High density lipoprotein (HDL-C) men < 40 mg/dL, women < 50 mg/dL
  * Blood pressure systolic ≥ 130 or diastolic ≥ 85 mmHg
  * Fasting glucose ≥ 100 mg/dL
Change in presence and severity of movement disorders | 0, 6 and 12 months
  Using SHRS and BARS (validated scales)
Change in brain volume | 0 and 12 months
  As measured with Magnetic Resonance Imaging (MRI)

OTHER OUTCOMES:
Change in immunological parameters | 0, 1 and 12 months
  * Multiplex immunoassay (including key cytokines, chemokines, metabolic markers, hormones, growth factors, acute phase reactants known to be associated with schizophrenia) will be measured at baseline.
  * Infectious disease profiling: (serology and the presence of specific infectious agents will be measured, including herpes simplex virus type-1 and -2, cytomegalovirus, Chlamydophila pneumonia, Chlamydophila psittaci and Toxoplasma Gondii) at baseline.
  * Flow cytometry (alterations in the number and functional responses of distinct sub-populations of blood cells will be analysed).
  * Selective reaction monitoring (a technique called SRM will be applied to investigate potential candidate biomarkers of drug response identified by proteome profiling [LC-MSE])
  * Gene expression and MicroRNA profiling (RNA expression of a set of 43 immune-related genes and miRNA-146a will be measured in total blood and monocytes isolated from PBMCs using Q-PCR).
Change in depressive symptoms | 0, 6 and 12 months
  Assessed with the Calgary Depression Scale for Schizophrenia (CDSS) total score
Number of participants with Adverse Events as a measure of safety and tolerability | 0 and 12 months
  Incidences (number and % of subjects with at least one occurrence) of key Serious Adverse Events (SAEs) and Adverse Events (AEs) will be presented per group.

CONTACTS AND LOCATIONS:
Overall Officials: Iris EC Sommer, Prof. dr., Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Derived] Zaki JK, Lago SG, Spadaro B, Rustogi N, Gangadin SS, Benacek J, Drexhage HA, de Witte LD, Kahn RS, Sommer IEC, Bahn S, Tomasik J. Exploring peripheral biomarkers of response to simvastatin supplementation in schizophrenia. Schizophr Res. 2024 Apr;266:66-74. doi: 10.1016/j.schres.2024.02.011. Epub 2024 Feb 19. PMID 38377869
- [Derived] Begemann MJH, Schutte MJL, van Dellen E, Abramovic L, Boks MP, van Haren NEM, Mandl RCW, Vinkers CH, Bohlken MM, Sommer IEC. Childhood trauma is associated with reduced frontal gray matter volume: a large transdiagnostic structural MRI study. Psychol Med. 2023 Feb;53(3):741-749. doi: 10.1017/S0033291721002087. Epub 2021 Jun 3. PMID 34078485
- [Derived] Begemann MJ, Schutte MJ, Slot MI, Doorduin J, Bakker PR, van Haren NE, Sommer IE. Simvastatin augmentation for recent-onset psychotic disorder: A study protocol. BBA Clin. 2015 Jul 3;4:52-58. doi: 10.1016/j.bbacli.2015.06.007. eCollection 2015 Dec. PMID 26674520